CLINICAL TRIAL: NCT00763620
Title: Assessment of the Diagnostic Capacity of a New Sampling Technique for Lower Respiratory Tract Culture for Patients With Acute Infectious Pneumonia Admitted in Intensive Care Unit and Non Intubated.
Brief Title: Assessment of the Diagnostic Capacity of the Mini-broncho Alveolar Lavage Performed Through a Suction Catheter
Acronym: Mini-LBA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: PLASTIMED Laboratory (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P080502
Record Dates: First submitted 2008-09-30; First posted 2008-10-01 (Estimated); Last update posted 2011-09-23 (Estimated); Status verified 2011-06

CONDITIONS: Bacterial Pneumonia
Keywords: Community acquired pneumonia; Nosocomial pneumonia; Mini bronchoalveolar lavage; Endotracheal aspirates; Expectorated sputum
MeSH Terms: conditions — Pneumonia, Bacterial; Community-Acquired Pneumonia; Healthcare-Associated Pneumonia | interventions — Catheters

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Catheter for mini bronchoalveolar lavage
  Interventions: Device: catheter for mini bronchoalveolar lavage

INTERVENTIONS:
Device: catheter for mini bronchoalveolar lavage — For each patient included an endotracheal aspiration and a mini bronchoalveolar lavage will be performed. After local anaesthesia, a suction catheter will be introduced in trachea by nasotracheal way. An endotracheal aspirate will be performed. Then, the mini bronchoalveolar lavage will be performed with the specific catheter introduced through the suction catheter. Expectorated sputum will also be ordered. This procedure will be performed once at the admission patient in intensive care unit.

SUMMARY:
The aim of this study is to develop a safe and effective technique to take sample for lower respiratory tract cultures easy to perform in conditions of acute respiratory failure and spontaneous ventilation for patients admitted in intensive care unit for acute infectious pneumonia and non intubated. The investigators perform sample collection with a mini bronchoalveolar lavage catheter introduced by nasotracheal way through a suction catheter. The purpose of the study is to assess the microbiological diagnostic capacity of this new technique.

DETAILED DESCRIPTION:
At the moment we lack an effective and safe technique to obtain lower respiratory tract cultures for patient with mild serious infectious pneumonia admitted in intensive care unit and non intubated. Invasive procedure may worsen respiratory distress and non invasive procedure such expectorated sputum culture is not enough effective. The purpose of the study is to assess the microbiological diagnosis capacity of a new technique for taking samples from the lower respiratory tract: mini bronchoalveolar lavage performed by naso tracheal way through a suction catheter.Each consecutive patient admitted in intensive care unit for a community acquired or nosocomial pneumonia and not requiring intubation and mechanical ventilation will be included. Written informed consent by patient himself will be required. For each patient, after the introduction of a suction catheter, an endotracheal aspiration will be performed. Then, the mini bronchoalveolar lavage will be performed through the suction catheter with a specific catheter.The whole time of the procedure is about ten minutes.Expectorated sputum will also be ordered for each patient.This study is a pilot and prospective study.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18
* Radiological diagnosis of pneumonia (community acquired or nosocomial)
* No microbiological diagnosis known
* Indication for culture of lower respiratory tract
* Admission in intensive care unit required

Exclusion Criteria:

* Age lower than 18
* Bronchospasm
* Coagulopathy ( Platelets count below 100 000/mm3, prothrombin time less than 50%, activated partial thromboplastin time ratio higher than 2)
* Intubation with mechanical ventilation
* Known microbiological diagnosis
* Incapacity for consenting himself to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2009-02; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure is the rate of positive microbiological culture | one year

SECONDARY OUTCOMES:
Comparison between rate of positive culture obtain with mini bronchoalveolar lavage and the two others techniques used in the sudy: endotracheal aspiration and expectorated sputum | one year
Feasibility of the procedure | ten minutes
The acceptance of the procedure | ten minutes
Physiological variables: heart and respiratory rate, oxygen saturation, blood pressure | before procedure and fifteen minutes after procedure
If applicable: complications of the procedure | one day
Time to obtain the result of the culture one day | one day
Time of the procedure | one day

CONTACTS AND LOCATIONS:
Overall Officials: Pascal MEYER, MD, Principal Investigator — Centre Hospitalier Sud Francilien - Corbeil Essonnes
Locations (1):
- Dr Pascal MEYER, Corbeil-Essonnes, Île-de-France Region, France

REFERENCES:
- [Derived] Meyer P, Rousseau H, Maillet JM, Thierry S, Sy O, Vicaut E, Thiolliere F, Choukroun G, Chergui K, Chevrel G, Maury E. Evaluation of blind nasotracheal suctioning and non-bronchoscopic mini-bronchoalveolar lavage in critically ill patients with infectious pneumonia: a preliminary study. Respir Care. 2014 Mar;59(3):345-52. doi: 10.4187/respcare.02356. Epub 2013 Jul 23. PMID 23882105